CLINICAL TRIAL: NCT01569451
Title: A Double Blinded, Randomized Study Comparing Rituximab Induction Therapy Followed by Glatiramer Acetate Therapy to Glatiramer Acetate Monotherapy in Patients With Relapsing Forms of Multiple Sclerosis
Brief Title: Comparison of Rituximab Induction Therapy Followed by Glatiramer Acetate
Acronym: GATEWAYII
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Rocky Mountain MS Research Group, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-1143
Record Dates: First submitted 2012-03-30; First posted 2012-04-03 (Estimated); Results first posted 2018-06-07 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Glatiramer Acetate; Rituximab; Relapsing forms of Multiple Sclerosis; Relapsing Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Rituximab; Glatiramer Acetate; Coat Protein Complex I

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- (Placebo and) Glatiramer Acetate (Active Comparator): Subjects will receive an intravenous (IV) infusion of placebo (normal saline) on study days 1 (baseline visit) and 15 according to the infusion protocol. On study day 28, all subjects will initiate standard Glatiramer Acetate therapy, 20 mg injected subcutaneously daily.
  Interventions: Drug: Glatiramer Acetate; Other: Placebo
- Rituximab and Glatiramer Acetate (R-GA) (Experimental): Subjects will receive an intravenous (IV) infusion of 1000 mg of rituximab on study days 1 (baseline visit) and 15 according to the rituximab infusion protocol. On study day 28, subjects will initiate standard Glatiramer Acetate therapy, 20 mg injected subcutaneously daily. There is no placebo arm.
  Interventions: Drug: Rituximab; Drug: Glatiramer Acetate

INTERVENTIONS:
Drug: Rituximab — intravenous (IV) infusion of 1000 mg of rituximab on study days 1 (baseline visit) and 15
  Other Names: Rituxan; MabThera
  Arms: Rituximab and Glatiramer Acetate (R-GA)
Drug: Glatiramer Acetate — 20 mg injected subcutaneously daily
  Other Names: Copolymer 1; Cop-1; Copaxone
Other: Placebo — Subjects will receive an intravenous (IV) infusion of 1000 mg of rituximab or placebo (normal saline) on study days 1 (baseline visit) and 15 according to the rituximab infusion protocol. On study day 28, all subjects will initiate standard GA therapy, 20 mg injected subcutaneously daily.
  Arms: (Placebo and) Glatiramer Acetate

SUMMARY:
The purpose of this study is (1) to determine if rituximab induction therapy followed by glatiramer acetate (GA) is substantially superior to placebo rituximab induction followed by GA for the treatment of clinically isolated syndrome (CIS) or relapsing forms of multiple sclerosis (RMS).

DETAILED DESCRIPTION:
This is a double blind, active comparator; single-center study involving up to 90 subjects with qualifying CIS or RMS. Subjects who are not screen-failures must be randomized within 60 days of signing the informed consent document. Subjects who are not randomized within these 60 days must be re-screened for enrollment into the study. Patients will be stratified based on their diagnosis of CIS or RMS (Relapsing Remitting or Secondary Progressive) and then randomly assigned at a 1:1 ratio to either rituximab induction followed by standard GA therapy (R-GA arm), or placebo induction followed by standard GA therapy (GA arm). Subjects will receive an intravenous (IV) infusion of 1000 mg of rituximab or placebo (normal saline) on study days 1 (baseline visit) and 15 according to the rituximab infusion protocol. On study day 28, all subjects will initiate standard GA therapy, 20 mg injected subcutaneously daily.

Study visits include screening, baseline/randomization (day 1), day 15, day 28 and then visits every 3 months for up to 2.5 years. A month is defined as 28 days. On study day 15, patients will receive the second dose of either rituximab or placebo; on study day 28 patients will begin treatment with GA therapy. Study days 15 and 28 have an acceptable window of +/- 4 days. Follow-up phone calls are conducted every month to assess adverse events and relapses. All monthly phone calls and quarterly visits must occur with a +/- 7 day window. Unscheduled office visits for the evaluation of symptoms suggestive of relapses will be scheduled as needed and may be prompted by questions elicited during the monthly safety and relapse assessment phone calls, or on the basis of a phone call initiated by the patient. In either case, those handling the phone call will interview the patient according to the questions described in the PDDS will be administered. If a subject reports new or worsening symptoms or there is a one point change in the PDDS score, an unscheduled visit will be necessary. The examining clinician will administer the Expanded Disability Status Scale (EDSS) but will be blinded to the PDDS score and type of visit (unscheduled or scheduled). The treating clinician will determine if the neurological change is considered a relapse based on EDSS scores provided by the EDSS evaluator and clinical presentation, and will make the decision whether or not corticosteroids should be administered for the treatment of a relapse. In addition, patients whose EDSS scores change sufficiently to qualify for SAD at either scheduled or unscheduled visits, will be asked to come in for an additional visit, 12 weeks later, to determine whether the change is sustained.

A sub-group of patients who provide informed consent will be enrolled in the Lumbar Puncture procedure. The procedure will be performed at the beginning of the study and at the 6 month visit. The objective will be to examine changes in CSF T and B cells and correlate them with evidence of disease activity by relapse, new MRI lesions and/or SAD. This procedure is optional for patients and will have no impact on the overall study. Patients who do decide to participate will sign an Addendum for Optional Procedure Consent Form The primary endpoint will be the number of disease-free patients, defined as patients without new lesions on brain MRI using the combined unique lesion approach (CUL), without sustained change in EDSS score over any 3-month period and without relapse. Once the last patient randomized has completed the final study visit for year 1 of the study, the data will be locked and an analysis performed on all data collected up to that point. An independent Data and Safety Monitoring Board (DSMB) will meet at initiation of the study and every 6 months thereafter until the end of the study. Members of the DSMB may unblind themselves at their discretion and the DSMB will include a statistician not directly involved in this study. If induction therapy fails to show superiority at any point, the study will be stopped.

Standardized brain MRIs with and without gadolinium contrast will be obtained at baseline, and month 6, 12, 18 and 24 months (for those patients reaching this point prior to the last enrolled patient reaching the 12 months follow-up visit) at UCD Anschutz Medical Campus. The treating clinician will have access to the MRI and can discuss the results openly with subjects. Standardized MRIs will be obtained and interpreted locally by a physician who will be blinded to the subject treatment to record the endpoints described above.

Assessments will be performed according to the schedule of events in section 4.1. Blinded examiners will be utilized for the EDSS, MSFC and low contrast visual acuity assessments. Lab results for B cell CD19+ counts will be collected by a blinded study coordinator who will have them reviewed on a monthly basis by a qualified member of the DSMB for safety assessment. But the CD19 B cell counts will not be available to the treating clinician unless needed for safety.

The treating clinician and the study coordinator will manage the clinical care and study related procedures. Complete metabolic panel (CMP) and liver function tests (LFT) will be obtained once a year as Standard of Care, or more often if deemed necessary by the treating clinician. Complete blood counts (CBC) with differential and CD19+ labs will be collected at Baseline, month 1 and every 3 months from baseline to monitor B cell recovery. The examining clinicians and primary study coordinator will be blinded to the CD19 lab results.

ELIGIBILITY:
Inclusion Criteria:

* 18 through 55 years of age
* Patients with CIS demonstrating one unifocal neurological event AND at least 2 T2-weighted brain lesions measuring a minimum of 6mm in diameter by MRI analysis; or a definite diagnosis of RMS, as defined by the 2005 revised McDonald criteria(1, 2), and have had at least one clinically defined relapse within the past year OR one GEL on an MRI within the past year
* Women of child-bearing potential must agree to practice an acceptable method of birth control
* No evidence of progressive multifocal leukoencephalopathy (PML) or primary central nervous system (PCNS) lymphoma
* Neurologically stable with no evidence of relapse or corticosteroid treatment within 30 days prior to randomization
* Subject must be able and willing to give meaningful, written informed consent prior to participation in the trial, in accordance with local regulatory requirements.

Exclusion Criteria:

* ≥ 15 GELs on baseline MRI
* Treatment with interferon β, natalizumab, or fingolimod within three months of randomization
* Treatment with mitoxantrone, cyclophosphamide, or any other chemotherapeutic agent for MS or malignancy within 12 months of randomization
* Attenuated live virus vaccination within 4 weeks of randomization
* Positive urine and serum pregnancy test at screening or baseline visit
* Any prior treatment with alemtuzumab or cladribine
* Unable to tolerate GA
* History of cardiac arrhythmias, angina or any other significant cardiac abnormalities
* History of clinically significant chronic disease of the immune system or a known immunodeficiency syndrome (HIV) other than MS
* White Blood Cell count of less than 2.5*10^9/L or lymphocyte count below 0.4*10^9/L
* Positive for any evidence of past, or current, hepatitis B and/or C infection
* History or presence of malignancy (except basal cell carcinoma)
* Clinically significant alcohol or drug abuse within past two years
* Any medical, psychiatric or other condition that could result in a subject not being able to give fully informed consent, or to comply with the protocol requirements
* Inability to undergo MRI scans or history of hypersensitivity to gadolinium- diethylenetriamine penta-acetic acid (DTPA)
* Participation in any clinical study evaluating another investigational drug or therapy within three months prior to randomization
* Any other condition that, in the Investigator's opinion, makes the subject unsuitable for participation in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2012-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Vollmer, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Honce JM, Nair KV, Sillau S, Valdez B, Miravalle A, Alvarez E, Schreiner T, Corboy JR, Vollmer TL. Rituximab vs placebo induction prior to glatiramer acetate monotherapy in multiple sclerosis. Neurology. 2019 Feb 12;92(7):e723-e732. doi: 10.1212/WNL.0000000000006916. Epub 2019 Jan 11. PMID 30635477

RESULTS

PARTICIPANT FLOW:
Groups:
- Glatiramer Acetate Therapy (GA): Subjects will receive an intravenous (IV) infusion of placebo (normal saline) on study days 1 (baseline visit) and 15 according to the infusion protocol. On study day 28, all subjects will initiate standard GA therapy, 20 mg injected subcutaneously daily.
  Glatiramer Acetate: 20 mg injected subcutaneously daily
- Rituximab + Glatiramer Acetate Therapy (R-GA): Subjects will receive an intravenous (IV) infusion of 1000 mg of rituximab on study days 1 (baseline visit) and 15 according to the rituximab infusion protocol. On study day 28, subjects will initiate standard GA therapy, 20 mg injected subcutaneously daily.
  Rituximab: intravenous (IV) infusion of 1000 mg of rituximab on study days 1 (baseline visit) and 15
  Glatiramer Acetate: 20 mg injected subcutaneously daily
Period: Overall Study
Arm/Group | Glatiramer Acetate Therapy (GA) | Rituximab + Glatiramer Acetate Therapy (R-GA)
Started | 26 | 27
Completed (Represents patients who completed the entire protocol. The analysis of key outcomes included 53) | 12 | 14
Not Completed | 14 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glatiramer Acetate Therapy (GA) | Rituximab + Glatiramer Acetate Therapy (R-GA) | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.64 (9.15) | 36.46 (8.31) | 36.55 (8.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 8 | 8 | 16
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 21 | 22 | 43
  Hispanic | 1 | 3 | 4
  Unknown | 4 | 2 | 6
Type of relapsing MS [Number; unit: participants]
  RRMS/SPMS | 24 | 25 | 49
  CIS | 2 | 2 | 4
Prior treatment with Tysabri [Number; unit: participants]
  Yes | 5 | 7 | 12
  No | 21 | 20 | 41
Prior treatment with Tysabri (within 6 months) [Number; unit: participants]
  Yes | 4 | 5 | 9
  No | 22 | 22 | 44
Expanded Disability Status Scale score at baseline [Mean (Standard Deviation); unit: units on a scale] — Physicians assess patients' cerebral, optic, brainstem, pyramidal, sensory, cerebellar, and bowel and bladder neurological symptoms. The physician then subjectively rates the patient on the ordinal EDSS scale. The EDSS scale emphasizes ambulatory ability. The EDSS scale ranges in half integer increments from 0.0 to 10.0. Larger numbers mean more disability, with 0.0 being everything normal and 10.0 being death due to MS.
  units on a scale | 2.63 (1.57) | 2.80 (1.78) | 2.72 (1.67)
Mean number of GEL at baseline [Mean (Standard Deviation); unit: lesions] | 0.54 (2.16) | 1.07 (2.53) | 0.81 (2.35)
Number with GEL at baseline [Number; unit: participants] | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Disease-free Patients
Description: Defined as patients without new lesions on brain MRI using the combined unique lesion approach (CUL), without sustained change in EDSS score over any 3-month period and without relapse. If a clear treatment effect is sustained in the R-GA arm, defined as a ≥ 70% decrease in brain lesions on MRI, using a CUL approach, attributable to MS and ≥ 70% reduction in annual relapse rates, compared to the GA arm, the study will continue under the extension protocol. If induction therapy fails to show superiority, at any point, the study will be stopped.
Time Frame: Baseline through 24 months
Population: Out to the last observation for each patient within 24 months (2 years) of follow up.
Measure: Number; unit: participants
Arm/Group | Glatiramer Acetate Therapy (GA) | Rituximab + Glatiramer Acetate Therapy (R-GA)
Number analyzed (Participants) | 26 | 27
participants | 5 | 12
Statistical Analysis 1: Comparison: Glatiramer Acetate Therapy (GA) vs Rituximab + Glatiramer Acetate Therapy (R-GA); Test type: Superiority or Other; p = 0.0493, Chi-squared

2. Secondary Outcome: Time to Treatment Failure
Description: Time itself is the outcome. Whenever treatment failure occurs for the first time within the follow up period of 24 months (2 years).
Time Frame: Baseline through 24 months
Population: Time itself is the outcome. Whenever treatment failure occurs for the first time within the follow up period of 24 months (2 years). Exposure time varies by patient. See exposure time outcome (post hoc).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Glatiramer Acetate Therapy (GA) | Rituximab + Glatiramer Acetate Therapy (R-GA)
Number analyzed (Participants) | 26 | 27
months | 11.29 [5.25 to 23.39] | 23.32 [14.64 to NA] — There was insufficient data to estimate the upper boundary of the confidence interval.
Statistical Analysis 1: Comparison: Glatiramer Acetate Therapy (GA) vs Rituximab + Glatiramer Acetate Therapy (R-GA); Test type: Superiority or Other; p = 0.0268, Peto

3. Secondary Outcome: Number of Subjects That Fail Treatment
Time Frame: Baseline through 24 months
Population: At any time within the follow up period of 24 months (2 years) out to the last observation.
Measure: Number; unit: participants
Arm/Group | Glatiramer Acetate Therapy (GA) | Rituximab + Glatiramer Acetate Therapy (R-GA)
Number analyzed (Participants) | 26 | 27
participants | 18 | 10
Statistical Analysis 1: Comparison: Glatiramer Acetate Therapy (GA) vs Rituximab + Glatiramer Acetate Therapy (R-GA); Test type: Superiority or Other; p = 0.0189, Chi-squared

4. Secondary Outcome: Number of Relapse-free Subjects
Description: Change in neurological symptoms in association with EDSS change is defined as relapse.
Time Frame: Baseline through 24 months
Population: Out to the last observation for each patient within 24 months (2 years) of follow up.
Measure: Number; unit: participants
Arm/Group | Glatiramer Acetate Therapy (GA) | Rituximab + Glatiramer Acetate Therapy (R-GA)
Number analyzed (Participants) | 26 | 27
participants | 17 | 21
Statistical Analysis 1: Comparison: Glatiramer Acetate Therapy (GA) vs Rituximab + Glatiramer Acetate Therapy (R-GA); Test type: Superiority or Other; p = 0.3167, Chi-squared

5. Secondary Outcome: Number of Patients Treated for Relapse With Corticosteroid
Time Frame: Baseline through 24 months
Population: At any time within the follow up period of 24 months (2 years) out to the last observation.
Measure: Number; unit: participants
Arm/Group | Glatiramer Acetate Therapy (GA) | Rituximab + Glatiramer Acetate Therapy (R-GA)
Number analyzed (Participants) | 26 | 27
participants | 9 | 4
Statistical Analysis 1: Comparison: Glatiramer Acetate Therapy (GA) vs Rituximab + Glatiramer Acetate Therapy (R-GA); Test type: Superiority or Other; p = 0.0940, Chi-squared

6. Secondary Outcome: Number of Subjects Who Experience Multiple Relapses
Time Frame: Baseline through 24 months
Population: At any time within the follow up period of 24 months (2 years) out to the last observation.
Measure: Number; unit: participants
Arm/Group | Glatiramer Acetate Therapy (GA) | Rituximab + Glatiramer Acetate Therapy (R-GA)
Number analyzed (Participants) | 26 | 27
participants | 3 | 1
Statistical Analysis 1: Comparison: Glatiramer Acetate Therapy (GA) vs Rituximab + Glatiramer Acetate Therapy (R-GA); Test type: Superiority or Other; p = 0.3507, Fisher Exact

7. Secondary Outcome: Number of Patients That Develop Sustained Accumulation of Disability
Description: Sustained accumulation of disability is defined as a 1 point change or more on the Expanded Disability Status Scale (EDSS); sustained for at least three months. Physicians assess patients' cerebral, optic, brainstem, pyramidal, sensory, cerebellar, and bowel and bladder neurological symptoms. The physician then subjectively rates the patient on the ordinal EDSS scale. The EDSS scale emphasizes ambulatory ability. The EDSS scale ranges in half integer increments from 0.0 to 10.0. Larger numbers mean more disability, with 0.0 being everything normal and 10.0 being death due to MS.
Time Frame: Baseline through 24 months
Population: At any observation within the follow up period of 24 months (2 years) out to the last observation.
Measure: Number; unit: participants
Arm/Group | Glatiramer Acetate Therapy (GA) | Rituximab + Glatiramer Acetate Therapy (R-GA)
Number analyzed (Participants) | 26 | 27
participants | 3 | 4
Statistical Analysis 1: Comparison: Glatiramer Acetate Therapy (GA) vs Rituximab + Glatiramer Acetate Therapy (R-GA); Test type: Superiority or Other; p = 1.0000, Fisher Exact

8. Secondary Outcome: Change From Baseline to 24 Months on the Multiple Sclerosis Functional Composite (MSFC) Z-score
Description: The MSFC consists of Timed 25 Foot Walk Tests, 9 Hole Peg Tests, and the Paced Auditory Serial Addition Test (PASAT), administered by clinicians. The subscales are then converted into Z-scores and averaged to create the MSFC Z-score. Larger values denote improvements.
Time Frame: Observations were recorded at baseline and 24 months.
Measure: Mean (95% Confidence Interval); unit: units on a scale (MSFC Z score)
Arm/Group | Glatiramer Acetate Therapy (GA) | Rituximab + Glatiramer Acetate Therapy (R-GA)
Number analyzed (Participants) | 25 | 26
units on a scale (MSFC Z score) | 0.5226 [-0.1840 to 1.2292] | 0.2630 [-0.0882 to 0.6141]
Statistical Analysis 1: Comparison: Glatiramer Acetate Therapy (GA) vs Rituximab + Glatiramer Acetate Therapy (R-GA); T-test; Test type: Superiority or Other; p = 0.4904, t-test, 2 sided

9. Secondary Outcome: Percentage of Subjects Worsening One Point or More on the Patient Determined Disease Steps (PDDS) Questionnaire
Description: For PDDS the patient selects an integer 0-8 according to their personal assessment of their degree of ambulatory disability. Larger numbers mean more disability, with 0 being no disability and 8 being bedridden. There is an unclassifiable category as well.
Time Frame: Baseline through 24 months
Population: At any time within the follow up period of 24 months (2 years) out to the last observation.
Measure: Count of Participants; unit: Participants
Arm/Group | Glatiramer Acetate Therapy (GA) | Rituximab + Glatiramer Acetate Therapy (R-GA)
Number analyzed (Participants) | 26 | 27
Participants | 6 | 9
Statistical Analysis 1: Comparison: Glatiramer Acetate Therapy (GA) vs Rituximab + Glatiramer Acetate Therapy (R-GA); Test type: Superiority or Other; p = 0.4073, Chi-squared

10. Secondary Outcome: Change in Mean Score on Performance Scales (Baseline to 24 Months)
Description: Performance scales measures patient assessments of disability in mobility (1-6), hand (1-5), vision (1-5), fatigue (1-5), cognitive (1-5), bladder and bowel, sensory (1-5), and spasticity (1-5). The overall measure of performance is the sum of subscales, ranging from 0 to 41. Larger numbers mean more disability, with 0 being no disability and the maximum number being total disability.
Time Frame: Baseline through 24 months
Population: At 24 months (2 years); the end of the study follow up period compared with baseline.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Glatiramer Acetate Therapy (GA) | Rituximab + Glatiramer Acetate Therapy (R-GA)
Number analyzed (Participants) | 26 | 27
units on a scale | 0.1466 [-1.4328 to 1.726] | 0.3477 [-1.6109 to 2.3062]
Statistical Analysis 1: Comparison: Glatiramer Acetate Therapy (GA) vs Rituximab + Glatiramer Acetate Therapy (R-GA); Test type: Superiority or Other; p = 0.8677, Mixed Models Analysis

11. Post Hoc Outcome: Exposure Time
Description: Values represent mean duration of treatment.
Time Frame: Measured in three month intervals from baseline to end of study.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | (Placebo and) Glatiramer Acetate | Rituximab and Glatiramer Acetate (R-GA)
Number analyzed (Participants) | 26 | 27
years | 1.517 (0.766) | 1.704 (0.830)
Statistical Analysis 1: Comparison: (Placebo and) Glatiramer Acetate vs Rituximab and Glatiramer Acetate (R-GA); Test type: Other — Mean difference between treatment groups; p = 0.3974, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Within 24 months (2 years) of follow up. Exposure time varied by patient.
Description: Out to the last observation for each patient within 24 months (2 years) of follow up. Exposure time varied by patient. See exposure time outcome (post hoc).
Arm/Group | Glatiramer Acetate Therapy (GA) | Rituximab + Glatiramer Acetate Therapy (R-GA)
Serious Adverse Events (participants affected / at risk) | 3/27 | 3/28
Other Adverse Events (participants affected / at risk) | 27/27 | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glatiramer Acetate Therapy (GA) (N=27) | Rituximab + Glatiramer Acetate Therapy (R-GA) (N=28)
Pulmonary (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
GI related (Gastrointestinal disorders) | 1 (1) | 0 (0)
Relapse related (Immune system disorders) | 1 (1) | 0 (0)
Neurological Condition (Nervous system disorders) | 1 (1) | 0 (0)
Other (General disorders) | 2 (2) | 2 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glatiramer Acetate Therapy (GA) (N=27) | Rituximab + Glatiramer Acetate Therapy (R-GA) (N=28)
Infusion-related reaction (General disorders) | 11 (13) | 19 (42)
Gastrointestinal Issues (Gastrointestinal disorders) | 7 (7) | 9 (15)
Influenza like illness (General disorders) | 13 (27) | 17 (28)
Injection site erythema (General disorders) | 2 (3) | 2 (2)
Fatigue (General disorders) | 10 (20) | 11 (35)
Injection-site reaction (General disorders) | 7 (11) | 8 (15)
URI (Infections and infestations) | 9 (12) | 8 (13)
UTI (Infections and infestations) | 6 (14) | 7 (13)
Bronchitis (Infections and infestations) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 10 (13) | 8 (11)
Depression (Psychiatric disorders) | 3 (5) | 5 (5)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 5 (6) | 7 (10)
Backpain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes